CLINICAL TRIAL: NCT05957042
Title: Pilot Study to Evaluate if Contrast Enhanced Ultrasound (CEUS) Can Predict Treatment Response in Triple Negative Breast Cancer (TNBC) Patients Receiving Combined Chemotherapy and Immune Checkpoint Inhibitors (ICI).
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Responsible Party left the institution and the study will not be started by other investigator
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Patton, Compliance Specialist-RQA, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22769
Record Dates: First submitted 2023-07-12; First posted 2023-07-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Contrast Enhanced Ultrasound
Keywords: Breast Cancer; Contrast Enhanced Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Evaluate whether CEUS can predict response on gold standard imaging in the same individuals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contrast Enhanced Ultrasound (with Lumason) (Experimental)
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — Up to 4.8mL administered intravenously

SUMMARY:
To find out if contrast enhanced ultrasound (CEUS) can be used to determine if patients receiving combined ICI therapy for triple negative breast cancer (TNBC) are responding to treatment earlier than standard of care MR or CT.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to sign and date the study-specific informed consent form.
* Stated willingness to comply with all study procedures and attend all study visits to the best of his or her ability for the duration of the study.
* Age greater than 18yo.
* Stage I-III TNBC or stage IV TNBC with intact breast primary.
* Planned combined ICI therapy as per SoC by treating oncologist.

Exclusion Criteria:

* Other clinical trials are not excluded but participation must be cleared with the other clinical trial PIs.
* Patients not suitable to undergo contrast enhanced ultrasound (i.e., pregnant women, known allergy to eggs, or a past allergic reaction to sonographic contrast or its components, such as polyethylene glycol (PEG))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Volume of mass on as visualized on contrast (Lumason) enhanced ultrasound at Baseline | Day 0 (Baseline)
Volume of mass on as visualized on contrast (Lumason) enhanced ultrasound at C2 | No later than week 5
Volume of mass on as visualized on contrast (Lumason) enhanced ultrasound at C3 | No later than week 9
Volume of mass on as visualized on contrast (Lumason) enhanced ultrasound at C4 | No later than week 13
Contrast (Lumason) enhanced ultrasound metric-area under the curve-at Baseline | Day 0 (Baseline)
Contrast (Lumason) enhanced ultrasound metric-area under the curve-at C2 | No later than week 5
Contrast (Lumason) enhanced ultrasound metric-area under the curve-at C3 | No later than week 9
Contrast (Lumason) enhanced ultrasound metric-area under the curve-at C4 | No later than week 13
Number of subjects who respond to treatment as reported on routine imaging. | No later than week 17

SECONDARY OUTCOMES:
Change in area under the curve (CEUS metric) between Baseline & C2 | No later than year 5
Change in area under the curve (CEUS metric) between Baseline & C3 | No later than year 5
Change in area under the curve (CEUS metric) between Baseline & C4 | No later than year 5
Change in area under the curve (CEUS metric) between C2 & C3 | No later than year 5
Change in area under the curve (CEUS metric) between C2 & C4 | No later than year 5
Change in area under the curve (CEUS metric) between C3 & C4 | No later than year 5
Number of subjects having pathologic complete response | No later than year 5
Overall survival (time to subject death) | No later than year 5

CONTACTS AND LOCATIONS:
Overall Officials: Seth Hardy, M.D., Principal Investigator — Assistant Professor - Department of Radiology, Penn State Health
Locations (1):
- Penn State Health College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No